CLINICAL TRIAL: NCT03487783
Title: A Multicenter, Randomized, Double-Blind, Flexible-Dosed, Placebo-Controlled, Parallel-Group Clinical Trial Evaluating the Efficacy and Safety of Aripiprazole Oral Solution in Children and Adolescents With Tourette's Syndrome
Brief Title: Aripiprazole Oral Solution in the Treatment of Children and Adolescents With Tourette's Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-403-00107
Record Dates: First submitted 2018-03-27; First posted 2018-04-04 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-01

CONDITIONS: Tourette Syndrome
Keywords: Tourette; Aripiprazole Oral Solution
MeSH Terms: conditions — Tourette Syndrome | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aripiprazole Oral Solution (Experimental): 1 mg/mL, 2-20 mg/day (2-20 mL/day), once daily for 8 weeks, administered at about the same time every day, either before or after meal
  Interventions: Drug: Aripiprazole Oral Solution
- Placebo Oral Solution (Placebo Comparator): 2-20 mg/day (2-20 mL/day), once daily for 8 weeks, administered at about the same time every day, either before or after meal
  Interventions: Drug: Placebo Oral Solution

INTERVENTIONS:
Drug: Aripiprazole Oral Solution — Aripiprazole 2-20 mg/day (2-20 mL/day)
  Other Names: Aripiprazole OS; Abilify
  Arms: Aripiprazole Oral Solution
Drug: Placebo Oral Solution — Placebo 2-20 mg/day (2-20 mL/day)
  Other Names: Placebo
  Arms: Placebo Oral Solution

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled trial designed to assess the safety, efficacy, tolerability and steady-state plasma trough concentration of flexible-dosed aripiprazole once-daily administration in children and adolescents with Tourette's syndrome. A total of around 120 subjects will be randomized to aripiprazole (2~20 mg) or placebo in a 1:1 ratio (approximately 60 subjects in each group), for treatment of 8 weeks.

DETAILED DESCRIPTION:
Screening phase: It can last up to 42 days, including the screening visit (V1), a washout period when applicable, additional screening visit (V1a) and baseline visit (V2). The screening phase will serve the following purposes: 1) To allow for appropriate washout of prohibited medications; 2) To review the screening data; 3) To establish a pretreatment baseline of critical outcome measures.

Treatment phase: It lasts 8 weeks; the purpose of the treatment phase is to assess the efficacy, safety, tolerability and steady-state plasma trough concentration of aripiprazole in the treatment of children and adolescents with Tourette's syndrome.

Safety follow-up phase: All subjects will be followed up for safety (adverse events) at Day 16 after the final medication via telephone

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent form must be obtained from a legal guardian (and the subject)
2. The subject and the designated guardian(s) or caregiver(s) are able to comprehend and satisfactorily comply with the protocol requirements, as evaluated by the investigator.
3. The subject is a male or female child or adolescent, 6-18 years of age (6≤ Age <18) at the time of Baseline Visit (V2);
4. The subject meets the current DSM-IV-TR diagnostic criteria for Tourette's syndrome and requires drug therapy;
5. The subject has a TTS ≥ 22 on the YGTSS at Baseline Visit (V2);

Exclusion Criteria:

1. Women of childbearing potential (WOCBP) who will not commit to utilizing the approved birth control methods or who will not remain abstinent during the trial and for 8 weeks following the final dose of study drug; Note: WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal [defined as amenorrhea 12 consecutive months; or women on hormone replacement therapy with documented serum follicle stimulating hormone level ≥ 35 mIU/mL].
2. Females who have a positive pregnancy test result or who are pregnant or breast-feeding;
3. Subjects who have secondary tic symptoms accompanied by late-onset tics, Huntington's chorea, neuroacanthocytosis, mental retardation, or autism;
4. Subjects who have comorbidities requiring drug therapy, such as attention deficit / attention-deficit hyperactivity, obsessive-compulsive disorder, or oppositional defiant disorder (if a case is judged by the investigator that drug therapy is not required for any of the above diseases during this study, then the patient is eligible to participate in this trial);
5. Subjects who have lower intelligence;
6. Subjects who have a current diagnosis of bipolar disorder, mental disorder, schizophrenia, or depressive disorder;
7. Subjects who have records of neuroleptic malignant syndrome;
8. Subjects who have experienced episodes of epileptic seizure in the past year;
9. Subjects who have a history of severe traumatic brain injury or stroke;
10. Subjects who have any unstable medical conditions or are currently ill (e.g., congenital heart disease, arrhythmia or cancer), which, in the investigator's judgment, will put them at a risk of major adverse event during this trial, or will interfere with safety and efficacy assessments
11. Subjects who require both drug therapy and cognitive-behavioral therapy (CBT, including habitual inversion therapy, cognitive therapy, relaxation training, etc.) during the trial period;
12. Patients with the following laboratory test results, vital signs, measurements, and electrocardiogram (ECG) results will be excluded:

    * QTc > 450 msec (male), QTc > 470 msec (female)
    * Platelets (< lower limit)
    * Hemoglobin (< lower limit)
    * Neutrophils (< lower limit)
    * AST (SGOT) or ALT (SGPT) (> upper limit)
    * Creatinine (> upper limit) Subjects should be excluded if they have any other abnormal laboratory tests, vital sign results, or ECG findings which in the investigator's judgment is medically significant and will impact the safety of the subject or the interpretation of the trial results;
13. Subjects who have a body weight of lower than 15 kg;
14. Subjects who have been known to be with allergy or hypersensitivity to aripiprazole or other dihydroquinolones (e.g., carteolol, vesnarinone and cilostazol);
15. Subjects who have participated in any clinical trial of any drugs within the past one month;
16. Subjects who may require concomitant treatments prohibited as per the protocol during the trial period (referring to Section 7 Prohibited and Restricted Therapies);
17. Subjects who were previously enrolled in clinical trials of aripiprazole (excluding investigator-sponsored trials);
18. Subjects who are considered to have developed resistance to antipsychotic drugs by the investigator due to lack of efficacy after receiving 2 different antipsychotic drugs at reasonable doses and at least 3 weeks of treatment with each respectively;
19. Subjects who are considered to have developed resistance to aripiprazole by the investigator due to lack of efficacy after an adequate time of treatment with adequate dose;

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline to Week 8 (or endpoint) in YGTSS TTS. | Baseline and 8 weeks (or endpoint)
  The objective of the primary analysis is to compare the efficacy of flexible-dosed aripiprazole oral solution (2~20 mg/day) with placebo in the suppression of tics in children and adolescents with a diagnosis of Tourette's syndrome. The efficacy is assessed by the changes of total tic scores (TTS) from randomization to the last visit (Week 8) on the Yale Global Tic Severity Scale (YGTSS).

SECONDARY OUTCOMES:
Percentage change from Baseline to Week 8 (or endpoint) in YGTSS TTS; | Baseline and 8 weeks (or endpoint)
  The efficacy is assessed by the percentage subjects changes of total tic scores (TTS) from randomization to the last visit (Week 8) on the Yale Global Tic Severity Scale (YGTSS)
Response rate on TS-CGI Improvement scale | Baseline and 8 weeks (or endpoint)
  The response rate (the percentage of patients with a score of 1 or 2) is assessed by TS-CGI Improvement scale from Baseline to Week 8 (or endpoint)
Partial remission rate on TS-CGI Improvement scale | Baseline and 8 weeks (or endpoint)
  The partial remission rate (the percentage of patients with a score of 3) is assessed by TS-CGI Improvement scale from Baseline to Week 8 (or endpoint)
Changes from Baseline to Week 8 (or endpoint) in TS-CGI Severity scale scores | Baseline and 8 weeks (or endpoint)
  The efficacy is assessed by changes from Baseline to Week 8 (or endpoint) in TS-CGI Severity scale scores

CONTACTS AND LOCATIONS:
Overall Officials: Patyman Juma, Study Director — Otsuka Beijing Research Institute
Locations (1):
- Beijing Anding Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He F, Luo J, Huang Y, Hao Y, Sun L, Ke X, Wu B, Chen Y, Han Y, Zhang Y, Liu J, Han H, Xian M, Uki M, Zheng Y. Randomized, double-blind, placebo-controlled trial of aripiprazole oral solution in children and adolescents with Tourette's disorder. Child Adolesc Psychiatry Ment Health. 2024 Jul 18;18(1):88. doi: 10.1186/s13034-024-00764-6. PMID 39026306